CLINICAL TRIAL: NCT03249350
Title: Experimental Mediation Research Aimed at Enhancing Adolescent Substance Abuse Treatment
Brief Title: Enhancing Adolescent Substance Abuse Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Social Learning Center (Other)
Responsible Party: Principal Investigator, Mike McCart, Senior Research Scientist, Oregon Social Learning Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01DA043578-01A1 (NIH)
Record Dates: First submitted 2017-08-10; First posted 2017-08-15 (Actual); Results first posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Substance Use Disorders
Keywords: Substance Use Disorders; Adolescents; Treatment; Mediation
MeSH Terms: conditions — Substance-Related Disorders; Negotiating

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Contingency Management (CM) (Active Comparator): This group will receive standard CM for adolescent substance abuse.
  Interventions: Behavioral: Standard Contingency Management (CM)
- Enhanced Contingency Management (CM+) (Experimental): This group will receive an enhanced CM protocol for adolescent substance abuse that targets parenting more intensely.
  Interventions: Behavioral: Enhanced Contingency Management (CM+)

INTERVENTIONS:
Behavioral: Standard Contingency Management (CM) — CM utilizes behavior modification & cognitive behavioral strategies to target adolescent substance use. Protocol components are as follows: (a) The provider introduces CM to the youth and caregiver and engages them in the intervention; (b) The provider conducts Antecedent-Behavior-Consequence (ABC) assessments of the youth's AOD use with the youth and caregiver; (c) Based on the results of the ABC assessments, self-management planning and drug refusal skills training are implemented by the provider in collaboration with the youth and caregiver; (d) Concurrently, a point and level system contract is established with the family, which provides the youth with rewards/privileges for negative drug and alcohol tests and disincentives (e.g., extra chores) for positive tests. Until continued abstinence is achieved, components "b" through "d" are repeated; (e) The provider collaborates with the family to develop plans for sustaining long-term abstinence. Typical duration of CM is 12-16 weeks.
  Arms: Standard Contingency Management (CM)
Behavioral: Enhanced Contingency Management (CM+) — The CM+ protocol adds the behavioral assessment and teaching system from Parent Management Training Oregon (PMTO) to standard CM to enhance parent's skill acquisition more intensely. PMTO's behavioral assessment and teaching system uses three processes to bring about changes in parenting: daily parent reports on youth behavior, anti-coercive problem-solving, and structured learning and in vivo practice of new parenting techniques.
  Arms: Enhanced Contingency Management (CM+)

SUMMARY:
The ultimate goal of this research is to facilitate rapid enhancement of youth substance abuse treatments by determining the key mechanisms of change (i.e., what to target more intensely to generate better outcomes). This work is critical because current outpatient adolescent substance abuse treatments yield only small to medium effects that diminish once treatment has ended. The proposed modern mediation study will address this serious public health problem by experimentally evaluating the most critical factors causing change in client outcomes during adolescent substance abuse treatment, directing the field to focus treatment efforts on those factors.

DETAILED DESCRIPTION:
Adolescents with substance use disorders (SUD) are at high risk for significant deleterious outcomes. Although several evidence-based practices for adolescent SUD exist, they yield only small to medium effects that rapidly diminish (30-70% 6-month relapse rates). A promising approach for determining how to enhance treatment is experimental mediation research. In contrast to traditional correlational mediation approaches, experimental mediation permits causal inference and is comprised of key steps: (A) Identify the putative mediating variable for a treatment. (B) Enhance the treatment to target that mediator more intensely. (C) Randomize youth to conditions, with the standard and enhanced versions of the treatment targeting different "levels" of the same mediator. (D) Measure the mediator and outcomes longitudinally. (E) Perform modern mediation analyses, coupled with analyses evaluating causal inference, to determine if changes in the mediator are responsible for changes in outcomes. This experimental test of mediation, focused on causality, facilitates rapid improvement of treatments by specifying change mechanisms to target in order to improve outcomes. These steps will be followed to elucidate the mediating processes in treatment for adolescent SUD, with the ultimate goal of enhancing the strength and durability of SUD treatments. The three most common putative mediating variables in adolescent SUD treatments are parent management, behavioral regulation, and peer relations. For this study, parent management was chosen as the target because it has evidenced the most potential for yielding generalizable change in youth outcomes and also has been shown to indirectly improve youths' behavioral regulation and peer relations. Of existing treatments for adolescent SUD, family-based Contingency Management (CM) was chosen as the treatment to enhance because it is highly amenable to an augmented focus on parenting, is less complex relative to other SUD treatments, and has amassed considerable support in terms of efficacy and dissemination potential. Thus, following experimental mediation steps, youth with SUD will be randomized to receive either standard CM or enhanced CM (i.e., CM+) that targets parenting more intensely. Repeated assessments for 12 months and longitudinal analyses will allow testing of mediating processes. The investigators will examine whether parent management skills mediate the effect of treatment on youth substance use and behavior problems (Aim 1). In addition, the investigators will determine whether parent management skills mediate the effect of treatment on youth behavioral regulation and deviant peer relations (Aim 2). Finally, the investigators will test whether behavioral regulation and deviant peer relations mediate the effect of parent management on youth substance use and behavior problems (Aim 3). Findings could have broad impact across multiple adolescent SUD treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 to 18 years
* Presence of current substance use disorder
* Availability of a parent/guardian willing to participate

Exclusion Criteria:

* Actively psychotic, suicidal, or homicidal
* Pervasive developmental disorder or metal retardation

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 129 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Adolescent and Family Clinic, OSLC Developments, Inc., Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study participants include adolescents aged 12-18 years with substance use disorders. All 129 adolescents enrolled in the study met the inclusion criteria and were randomized to treatment. Only adolescents were considered enrolled in the study.
Period: Overall Study
Arm/Group | Standard Contingency Management (CM) | Enhanced Contingency Management (CM+)
Started | 66 | 63
Completed | 61 | 55
Not Completed | 5 | 8
Not completed — Participant did not initiate treatment | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Contingency Management (CM) | Enhanced Contingency Management (CM+) | Total
Number analyzed (Participants) | 66 | 63 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.76 (1.49) | 14.98 (1.36) | 14.87 (1.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 26 | 50
  Male | 42 | 37 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 16 | 24
  Not Hispanic or Latino | 57 | 47 | 104
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 1 | 2 | 3
  White | 58 | 52 | 110
  More than one race | 1 | 4 | 5
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 66 | 63 | 129
Total Positive Urine Drug Screen [Mean (Standard Deviation); unit: count of positive screens] — The total number of substances a participant tested positive for at their baseline urine drug screen.
  count of positive screens | 0.82 (0.72) | 0.84 (0.65) | 0.83 (0.69)
Any Positive Urine Drug Screen [Number; unit: proportion of participants] — A 10-panel urine screen was collected from each adolescent at baseline. Each adolescent was scored as a 1 or a 0, where 1 indicates they tested positive for any substance on their baseline urine screen and 0 indicates they didn't test positive for any substances on their baseline urine screen. Numbers represent the proportion of participants with a positive screen result at baseline.
  proportion of participants | 0.68 | 0.73 | 0.71
Global Appraisal of Individual Needs (GAIN) Substance Problem [Mean (Standard Deviation); unit: units on a scale] — The Global Appraisal of Individual Needs (GAIN) Substance Problems Subscale measures the presence of each DSM-V criterion for a substance use disorder and lower severity symptoms. Scores range from 0 to 16, where higher scores indicate the presence of more criterion/symptoms.
  units on a scale | 6.73 (4.33) | 7.19 (4.73) | 6.95 (4.52)
Global Appraisal of Individual Needs (GAIN) Substance Dependence [Mean (Standard Deviation); unit: units on a scale] — The Global Appraisal of Individual Needs (GAIN) Substance Dependence Subscale measures the number of dependence related symptoms. Scores range from 0 to 7, where higher scores indicate the presence of more symptoms.
  units on a scale | 3.15 (2.33) | 3.27 (2.49) | 3.21 (2.4)
Global Appraisal of Individual Needs (GAIN) Substance Frequency [Mean (Standard Deviation); unit: units on a scale] — The Global Appraisal of Individual Needs (GAIN) Frequency Subscale measures the frequency of substance use of 16 different substances over the past 30 days. Scores range from 0 to 100, where higher scores indicate higher frequency use.
  units on a scale | 22.89 (17.37) | 21.9 (17.42) | 22.4 (17.3)
Child Behavior Checklist (CBCL) - Externalizing Youth Report [Mean (Standard Deviation); unit: units on a scale] — This is a 35-item Subscale of the Child Behavior Checklist (CBCL) measuring externalizing behaviors from the youth's self-report. It assesses outward-directed behaviors such as aggression, defiance, hyperactivity, and rule-breaking. Scores range from 0 to 70, where higher scores indicate the presence of more externalizing behavior problems.
  units on a scale | 22.88 (10.19) | 24.6 (11.09) | 23.72 (10.63)
Child Behavior Checklist (CBCL) - Externalizing Parent Report [Mean (Standard Deviation); unit: units on a scale] — This is a 35-item subscale of the Child Behavior Checklist (CBCL) measuring externalizing behaviors from the parent's report on youth's behaviors. It assesses outward-directed behaviors such as aggression, defiance, hyperactivity, and rule-breaking. Scores range from 0 to 70, where higher scores indicate the presence of more externalizing behavior problems.
  units on a scale | 31.95 (15.18) | 28.03 (13.91) | 30.04 (14.65)
Peer Delinquency [Mean (Standard Deviation); unit: units on a scale] — The Peer Delinquency Scale of the Pittsburgh Youth Study Interview comprises 20 questions rated on a 4-point scale (0 = none to 4 = all) concerning the proportion of friends of the subject that have engaged in a variety of antisocial and delinquent behaviors over the past 30 days. Scores range from 0 to 80, where higher scores indicate a higher proportion of delinquent friends.
  units on a scale | 15.42 (13.75) | 14.83 (10.74) | 15.13 (12.33)
Positive Peer Activity - Youth Report [Mean (Standard Deviation); unit: units on a scale] — The Positive Peer Activity Scale of the Pittsburgh Youth Study Interview comprises 10 questions rated on a 4-point scale (0 = none to 4 = all) concerning the proportion of friends of the subject that have engaged in a variety of prosocial activities over the past 30 days. Scores range from 0 to 40, where higher scores indicate a higher proportion of prosocial friends. This is measured from the youth's self-report.
  units on a scale | 16.62 (5.92) | 15.16 (5.94) | 15.91 (12.33)
Positive Peer Activity - Parent Report [Mean (Standard Deviation); unit: units on a scale] — The Positive Peer Activity Scale of the Pittsburgh Youth Study Interview comprises 10 questions rated on a 4-point scale (0 = none to 4 = all) concerning the proportion of friends of the subject that have engaged in a variety of prosocial activities over the past 30 days. Scores range from 0 to 40, where higher scores indicate a higher proportion of prosocial friends. This is measured from the parent's report on youth's friends.
  units on a scale | 9.8 (5.29) | 10.51 (6.56) | 10.15 (5.93)
Alabama Parenting Questionnaire (APQ) Involvement - Youth [Mean (Standard Deviation); unit: units on a scale] — A 10-item subscale of the Alabama Parenting Questionnaire (APQ) that assesses the extent of a parent's engagement in their child's life through shared activities and emotional support. Higher scores indicate greater parental engagement in the child's life. Scores range from 10-50. High scores suggest strong emotional and practical involvement, which is generally protective against behavioral problems.This is measured through youths' reports on parents' behaviors.
  units on a scale | 30.53 (7.38) | 30.79 (6.58) | 30.66 (6.98)
Alabama Parenting Questionnaire (APQ) Positive Parenting - Youth [Mean (Standard Deviation); unit: units on a scale] — A 6-item subscale of the Alabama Parenting Questionnaire (APQ) that measures positive parenting through the frequency of praise and reinforcement. Scores range from 6 -30. High scores reflect the frequent use of praise and rewards, which are associated with better child compliance and emotional well-being. This is measured through youths' reports on parents' behaviors.
  units on a scale | 19.82 (4.89) | 19.57 (4.51) | 19.7 (4.69)
Alabama Parenting Questionnaire (APQ) Poor Monitoring - Youth [Mean (Standard Deviation); unit: units on a scale] — A 10-item subscale of the Alabama Parenting Questionnaire (APQ) that measures parents' monitoring and supervision of their child's activities and whereabouts. Scores range from 10-50. Higher scores indicate less parental awareness of the child's activities. Elevated scores are associated with an increased risk of delinquency and externalizing behaviors. This is measured through youths' reports on parents' behaviors.
  units on a scale | 25.15 (6.42) | 24.63 (6.38) | 24.9 (6.38)
Alabama Parenting Questionnaire (APQ) Inconsistent Discipline- Youth [Mean (Standard Deviation); unit: units on a scale] — A 6-item subscale of the Alabama Parenting Questionnaire (APQ) that measures parents' discipline activity and the variability in rule enforcement and consequences. Scores range from 6 -30. High scores suggest unpredictable enforcement of rules, which can undermine authority and increase behavioral issues. This is measured through youths' reports on parents' behaviors.
  units on a scale | 14.8 (5.07) | 14.6 (4.48) | 14.71 (4.77)
Alabama Parenting Questionnaire (APQ) Corporal Punishment - Youth [Mean (Standard Deviation); unit: units on a scale] — A 3-item subscale of the Alabama Parenting Questionnaire (APQ) that measures parents' use of corporal punishment or physical discipline. Scores range from 3-15. Higher scores may indicate reliance on punitive strategies, which are associated with negative child outcomes such as aggression. This is measured through youths' reports on parents' behaviors.
  units on a scale | 5.11 (1.84) | 5.43 (1.54) | 5.26 (1.7)
Alabama Parenting Questionnaire (APQ) Involvement - Parent [Mean (Standard Deviation); unit: units on a scale] — A 10-item subscale of the Alabama Parenting Questionnaire (APQ) that assesses the extent of a parent's engagement in their child's life through shared activities and emotional support. Higher scores indicate greater parental engagement in the child's life. Scores range from 10-50. High scores suggest strong emotional and practical involvement, which is generally protective against behavioral problems. This is measured through parents' self-reports of their own behaviors.
  units on a scale | 24.85 (4.89) | 25.46 (5.13) | 25.15 (5)
Alabama Parenting Questionnaire (APQ) Positive Parenting - Parent [Mean (Standard Deviation); unit: units on a scale] — A 6-item subscale of the Alabama Parenting Questionnaire (APQ) that measures positive parenting through the frequency of praise and reinforcement. Scores range from 6-30. High scores reflect the frequent use of praise and rewards, which are associated with better child compliance and emotional well-being. This is measured through parents' self-reports of their own behaviors.
  units on a scale | 18.09 (3.28) | 17.16 (3.69) | 17.64 (3.5)
Alabama Parenting Questionnaire (APQ) Poor Monitoring - Parent [Mean (Standard Deviation); unit: units on a scale] — A 10-item subscale of the Alabama Parenting Questionnaire (APQ) that measures parents' monitoring and supervision of their child's activities and whereabouts. Scores range from 10-50. Higher scores indicate less parental awareness of the child's activities. Elevated scores are associated with an increased risk of delinquency and externalizing behaviors. This is measured through parents' self-reports of their own behaviors.
  units on a scale | 14.35 (6.26) | 14.89 (6.48) | 14.61 (6.35)
Alabama Parenting Questionnaire (APQ) Inconsistent Discipline- Parent [Mean (Standard Deviation); unit: units on a scale] — A 6-item subscale of the Alabama Parenting Questionnaire (APQ) that measures parents' discipline activity and the variability in rule enforcement and consequences. Scores range from 6-30. High scores suggest unpredictable enforcement of rules, which can undermine authority and increase behavioral issues. This is measured through parents' self-reports of their own behaviors.
  units on a scale | 10.09 (4.6) | 10.62 (4.03) | 10.35 (4.32)
Alabama Parenting Questionnaire (APQ) Corporal Punishment - Parent [Mean (Standard Deviation); unit: units on a scale] — A 3-item subscale of the Alabama Parenting Questionnaire (APQ) that measures parents' use of corporal punishment or physical discipline. Scores range from 3-15. Higher scores may indicate reliance on punitive strategies, which are associated with negative child outcomes such as aggression. This is measured through parents' self-reports of their own behaviors.
  units on a scale | 1.95 (1.34) | 2.11 (1.25) | 2.03 (1.29)
Early Adolescent Temperament Questionnaire (EATQ) Effortful Control Factor - Youth [Mean (Standard Deviation); unit: units on a scale] — Youth report of youth inhibitory control as assessed by the mean score on the Effortful Control factor from the Early Adolescent Temperament Questionnaire. Scores on individual items and factor range from 1=Very false to 5=Very true. Higher scores equal higher youth effortful control.
  units on a scale | 2.96 (0.63) | 2.8 (0.53) | 2.88 (0.59)
Early Adolescent Temperament Questionnaire (EATQ) Effortful Control Factor - Parent [Mean (Standard Deviation); unit: units on a scale] — Parent report of youth inhibitory control as assessed by the mean score on the Effortful Control factor from the Early Adolescent Temperament Questionnaire. Scores on individual items and factor range from 1=Very false to 5=Very true. Higher scores equal higher youth effortful control.
  units on a scale | 2.4 (0.6) | 2.44 (0.54) | 2.42 (0.57)
Go-No-Go Percent Correct [Mean (Standard Deviation); unit: percent correct] — Youth performance of youth inhibitory control as assessed by the percent correct on no go trials on computerized go/no-go task.
  percent correct | 0.74 (0.15) | 0.74 (0.15) | 0.74 (0.15)
Behavioral Inhibition and Behavioral Activation Systems (BIS-BAS) Drive - Youth [Mean (Standard Deviation); unit: units on a scale] — Youth report of youth risk taking as assessed by the sum score on the Drive subscale from the Behavioral Inhibition System and Behavioral Activation System scales. Scores on individual items and subscale range from 1=Strongly agree to 4=Strongly disagree and scores range from 4 to 16. Higher scores equal higher youth behavioral activation (drive).
  units on a scale | 11.3 (2.41) | 11.19 (2.31) | 11.25 (2.36)
Behavioral Inhibition and Behavioral Activation Systems (BIS-BAS) Fun Seeking - Youth [Mean (Standard Deviation); unit: units on a scale] — Youth report of youth risk taking as assessed by the sum score on the Fun Seeking subscale from the Behavioral Inhibition System and Behavioral Activation System scales. Scores on individual items and subscale range from 1=Strongly agree to 4=Strongly disagree and scores range from 4 to 16. Higher scores equal higher youth behavioral activation (fun seeking).
  units on a scale | 11.86 (1.8) | 12.46 (1.92) | 12.16 (1.88)
Behavioral Inhibition and Behavioral Activation Systems (BIS-BAS) Reward Responsiveness - Youth [Mean (Standard Deviation); unit: units on a scale] — Youth report of youth risk taking as assessed by the sum score on the Reward Responsiveness subscale from the Behavioral Inhibition System and Behavioral Activation System. Scores on individual items and subscale range from 1=Strongly agree to 4=Strongly disagree and scores range from 5 to 20. Higher scores equal higher youth behavioral activation (reward responsiveness).
  units on a scale | 15.35 (2.43) | 15.41 (2.32) | 15.38 (2.37)
Behavioral Inhibition and Behavioral Activation Systems (BIS-BAS) Drive - Parent [Mean (Standard Deviation); unit: units on a scale] — Parent report of youth risk taking as assessed by the sum score on the Drive subscale from the Behavioral Inhibition System and Behavioral Activation System scales. Scores on individual items and subscale range from 1=Strongly agree to 4=Strongly disagree and scores range from 4 to 16. Higher scores equal higher youth behavioral activation (drive).
  units on a scale | 11.91 (2.05) | 11.44 (2.6) | 11.68 (2.34)
Behavioral Inhibition and Behavioral Activation Systems (BIS-BAS) Fun Seeking - Parent [Mean (Standard Deviation); unit: units on a scale] — Parent report of youth risk taking as assessed by the sum score on the Fun Seeking subscale from the Behavioral Inhibition System and Behavioral Activation System scales. Scores on individual items and subscale range from 1=Strongly agree to 4=Strongly disagree and scores range from 4 to 16. Higher scores equal higher youth behavioral activation (fun seeking).
  units on a scale | 12 (1.72) | 11.84 (1.95) | 11.92 (1.83)
Behavioral Inhibition and Behavioral Activation Systems (BIS-BAS) Reward Responsiveness - Parent [Mean (Standard Deviation); unit: units on a scale] — Parent report of youth risk taking as assessed by the sum score on the Reward Responsiveness subscale from the Behavioral Inhibition System and Behavioral Activation System scales. Scores on individual items and subscale range from 1=Strongly agree to 4=Strongly disagree and scores range from 5 to 20. Higher scores equal higher youth behavioral activation (reward responsiveness).
  units on a scale | 15.47 (2.19) | 15.03 (2.36) | 15.26 (2.28)
Balloon Analog Risk Task (BART) Number of Pumps [Mean (Standard Deviation); unit: pumps] — Youth performance on computerized Balloon Analogue Risk Task (automatic version) that requires participants to enter the number of times that they want to pump to inflate a computer-generated balloon, with participants earning a point for each pump but losing all of the points if the balloon pops before the selected number of pumps. The mean number of pumps on all trials is reported. Scores range from 0 to 126. Higher scores equal higher youth risk taking behavior.
  pumps | 48.49 (12.17) | 51.72 (13.33) | 50.05 (12.79)

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline Scores Compared to Post-Treatment Scores, Any Positive Youth Urine Drug/Alcohol Screens (Measured at 0, 2, 4, 6, 9, & 12 Months).
Description: Any positive urine screens for tetrahydrocannabinol (THC), synthetic THC, amphetamines, opiates, phencyclidine (PCP), cocaine, and/or alcohol metabolites (ethyl glucuronide, ethyl sulfate).
Time Frame: Baseline to 12 months
Measure: Mean (Standard Error); unit: positive test per timepoint
Arm/Group | Standard Contingency Management (CM) | Enhanced Contingency Management (CM+)
Number analyzed (Participants) | 66 | 63
positive test per timepoint
  Baseline timepoint | 0.68 (0.47) | 0.73 (0.45)
  2 months | 0.60 (0.49) | 0.55 (0.50)
  4 months | 0.51 (0.51) | 0.41 (0.50)
  6 months | 0.50 (0.51) | 0.54 (0.51)
  9 months | 0.53 (0.51) | 0.37 (0.49)
  12 months | 0.44 (0.50) | 0.45 (0.51)
Statistical Analysis 1: Comparison: Standard Contingency Management (CM) vs Enhanced Contingency Management (CM+); Mixed effects regression model tested for between-group differences in change over time; Test type: Superiority; p = 0.49, Mixed Models Analysis; Slope = -0.05, Standard Error of Mean 0.07

2. Secondary Outcome: Changes From Baseline Scores Compared to Post-Treatment Scores for Youth Problem Behaviors (Measured at 0, 2, 4, 6, 9, & 12 Months).
Description: Youth problem behaviors as measured by the Child Behavior Checklist (parent-report) and the Youth Self Report.
  This is a 35-item Subscale of the Child Behavior Checklist (CBCL) measuring externalizing behaviors from the youth's self-report. It assesses outward-directed behaviors such as aggression, defiance, hyperactivity, and rule-breaking. Scores range from 0 to 70, where higher scores indicate the presence of more externalizing behavior problems.
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Contingency Management (CM) | Enhanced Contingency Management (CM+)
Number analyzed (Participants) | 66 | 63
score on a scale
  Baseline | 22.88 (10.19) | 24.6 (11.09)
  2 Months | 18.07 (11.09) | 19.15 (10.35)
  4 Months | 17.05 (9.94) | 16.53 (11.23)
  6 Months | 16.26 (8.97) | 15.06 (9.79)
  9 Months | 16.06 (9.02) | 13.59 (11.45)
  12 Months | 15.82 (10.89) | 14.4 (11.07)
Statistical Analysis 1: Comparison: Standard Contingency Management (CM) vs Enhanced Contingency Management (CM+); Mixed effects regression model tested for between-group differences in change over time; Test type: Superiority; p = 0.92, Mixed Models Analysis; Slope = 0.02, Standard Error of Mean 0.19

3. Secondary Outcome: Youth Receipt of Required Contingency Management (CM) Treatment Components.
Description: All treatment sessions were audio-recorded. A random selection of tapes was coded by trained raters to indicate the presence or absence of CM treatment components. Scores on this outcome reflect the proportion of components delivered, with higher scores indicating the presence of more treatment components.
Time Frame: Course of treatment (length varied by participant)
Measure: Mean (Standard Error); unit: proportion of components received
Arm/Group | Standard Contingency Management (CM) | Enhanced Contingency Management (CM+)
Number analyzed (Participants) | 66 | 63
proportion of components received
  Cognitive Behavioral Components | 0.16 (0.01) | 0.11 (0.01)
  Behavioral Modification Components | 0.33 (0.01) | 0.37 (0.01)
Statistical Analysis 1: Comparison: Standard Contingency Management (CM) vs Enhanced Contingency Management (CM+); Cognitive Behavioral Components; Test type: Superiority; p < 0.001, ANOVA; Main effect of group, F=13.58
Statistical Analysis 2: Comparison: Standard Contingency Management (CM) vs Enhanced Contingency Management (CM+); Behavioral Modification Components; Test type: Superiority; p = 0.08, ANOVA; Main effect of group, F=3.02

4. Secondary Outcome: Changes From Baseline Scores Compared to Post-Treatment Scores for Parent Management - Inconsistent Discipline Subscale - Parent Report(Measured at 0, 2, 4, 6, 9, & 12 Months).
Description: A 6-item subscale of the Alabama Parenting Questionnaire (APQ) that measures parents' discipline activity and the variability in rule enforcement and consequences. Scores range from 6-30. High scores suggest unpredictable enforcement of rules, which can undermine authority and increase behavioral issues. This is measured through parents' self-reports of their own behaviors.
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Contingency Management (CM) | Enhanced Contingency Management (CM+)
Number analyzed (Participants) | 66 | 63
score on a scale
  Baseline - Parent | 10.09 (4.6) | 10.62 (4.03)
  2 months - Parent | 9.63 (4.08) | 9.27 (3.59)
  4 months - Parent | 9.7 (4.93) | 9.11 (4.37)
  6 months - Parent | 9.55 (4.52) | 7.93 (3.67)
  9 months - Parent | 8.07 (4.52) | 7.56 (3.91)
  12 months - Parent | 9.48 (4.27) | 7.4 (3.83)
Statistical Analysis 1: Comparison: Standard Contingency Management (CM) vs Enhanced Contingency Management (CM+); Mixed effects regression model tested for between-group differences in change over time; Test type: Superiority; p = 0.09, Mixed Models Analysis; Slope = -0.11, Standard Error of Mean 0.07

5. Secondary Outcome: Changes From Baseline Scores Compared to Post-Treatment Scores for Parent Management - Positive Parenting Subscale - Parent Report (Measured at 0, 2, 4, 6, 9, & 12 Months).
Description: A 6-item subscale of the Alabama Parenting Questionnaire (APQ) that measures positive parenting through the frequency of praise and reinforcement. Scores range from 6-30. High scores reflect the frequent use of praise and rewards, which are associated with better child compliance and emotional well-being. This is measured through parents' self-reports of their own behaviors.
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Standard Contingency Management (CM) | Enhanced Contingency Management (CM+)
Number analyzed (Participants) | 66 | 63
Scores on a scale
  Baseline - Parent | 18.09 (3.28) | 17.16 (3.69)
  2 months - Parent | 18.27 (3.72) | 17.06 (3.62)
  4 months - Parent | 17.66 (4.02) | 17.48 (3.17)
  6 months - Parent | 18.45 (3.85) | 18.05 (3.22)
  9 months - Parent | 18.22 (3.99) | 18.15 (3.52)
  12 months - Parent | 18.55 (3.27) | 18.14 (4.27)
Statistical Analysis 1: Comparison: Standard Contingency Management (CM) vs Enhanced Contingency Management (CM+); Mixed effects regression model tested for between-group differences in change over time; Test type: Superiority; p = 0.95, Mixed Models Analysis; Slope = -0.004, Standard Error of Mean 0.06

6. Secondary Outcome: Changes From Baseline Scores Compared to Post-Treatment Scores for Parent Management - Poor Monitoring Subscale - Parent Report (Measured at 0, 2, 4, 6, 9, & 12 Months).
Description: Parent management practices as measured by the Alabama Parenting Questionnaire (APQ) (parent-report).
  A 10-item subscale of the Alabama Parenting Questionnaire (APQ) that measures parents' monitoring and supervision of their child's activities and whereabouts. Scores range from 10-50. Higher scores indicate less parental awareness of the child's activities. Elevated scores are associated with an increased risk of delinquency and externalizing behaviors. This is measured through parents' self-reports of their own behaviors.
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Contingency Management (CM) | Enhanced Contingency Management (CM+)
Number analyzed (Participants) | 66 | 63
score on a scale
  Baseline - Parent | 14.35 (6.26) | 14.89 (6.48)
  2 months - Parent | 14.29 (5.96) | 14.73 (7.28)
  4 months - Parent | 13.59 (6.69) | 14.3 (7.39)
  6 months - Parent | 13.6 (7.44) | 13.02 (6.02)
  9 months - Parent | 11.83 (6.01) | 12.03 (6.27)
  12 months - Parent | 13.09 (7.07) | 12.69 (6.92)
Statistical Analysis 1: Comparison: Standard Contingency Management (CM) vs Enhanced Contingency Management (CM+); APQ - Poor Monitoring - Parent Report Mixed effects regression model tested for between-group differences in change over time; Test type: Superiority; p = 0.88, Mixed Models Analysis; Slope = 0.02, Standard Error of Mean 0.11

7. Secondary Outcome: Changes From Baseline Scores Compared to Post-Treatment Scores for Parent Management - Inconsistent Discipline Subscale (Youth Report) (Measured at 0, 2, 4, 6, 9, & 12 Months).
Description: A 6-item subscale of the Alabama Parenting Questionnaire (APQ) that measures parents' discipline activity and the variability in rule enforcement and consequences. Scores range from 6 -30. High scores suggest unpredictable enforcement of rules, which can undermine authority and increase behavioral issues. This is measured through youths' reports on parents' behaviors.
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Contingency Management (CM) | Enhanced Contingency Management (CM+)
Number analyzed (Participants) | 66 | 63
score on a scale
  Baseline - Youth | 14.8 (5.07) | 14.6 (4.48)
  2 months - Youth | 14.37 (4.56) | 13.63 (4.28)
  4 months - Youth | 13.58 (4.92) | 13.56 (3.47)
  6 months - Youth | 13.09 (4.75) | 12.65 (4.12)
  9 months - Youth | 12.74 (5.24) | 13.09 (3.87)
  12 months - Youth | 13.19 (5.59) | 12.69 (3.49)
Statistical Analysis 1: Comparison: Standard Contingency Management (CM) vs Enhanced Contingency Management (CM+); Mixed effects regression model tested for between-group differences in change over time; Test type: Superiority; p = 0.06, Mixed Models Analysis; Slope = 0.16, Standard Error of Mean 0.09

8. Secondary Outcome: Changes From Baseline Scores Compared to Post-Treatment Scores for Parent Management - Positive Parenting Subscale - Youth Report (Measured at 0, 2, 4, 6, 9, & 12 Months).
Description: A 6-item subscale of the Alabama Parenting Questionnaire (APQ) that measures positive parenting through the frequency of praise and reinforcement. Scores range from 6-30. High scores reflect the frequent use of praise and rewards, which are associated with better child compliance and emotional well-being. This is measured through youths' report on parents' behaviors.
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Contingency Management (CM) | Enhanced Contingency Management (CM+)
Number analyzed (Participants) | 66 | 63
score on a scale
  Baseline - Youth | 19.82 (4.89) | 19.57 (4.51)
  2 months - Youth | 18.93 (5.32) | 19.59 (5.36)
  4 months - Youth | 19.85 (5.09) | 19.41 (4.63)
  6 months - Youth | 19.83 (5.48) | 19.79 (5.08)
  9 months - Youth | 19.26 (5.68) | 20.13 (5.45)
  12 months - Youth | 19.19 (5.39) | 19.69 (5.28)
Statistical Analysis 1: Comparison: Standard Contingency Management (CM) vs Enhanced Contingency Management (CM+); Mixed effects regression model tested for between-group differences in change over time; Test type: Superiority; p = 0.50, Mixed Models Analysis; Slope = -0.06, Standard Error of Mean 0.09

9. Secondary Outcome: Changes From Baseline Scores Compared to Post-Treatment Scores for Parent Management - Poor Monitoring Subscale - Youth Report (Measured at 0, 2, 4, 6, 9, & 12 Months).
Description: A 10-item subscale of the Alabama Parenting Questionnaire (APQ) that measures parents' monitoring and supervision of their child's activities and whereabouts. Scores range from 10-50. Higher scores indicate less parental awareness of the child's activities. Elevated scores are associated with an increased risk of delinquency and externalizing behaviors. This is measured through youths' reports on parents' behaviors.
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Contingency Management (CM) | Enhanced Contingency Management (CM+)
Number analyzed (Participants) | 66 | 63
score on a scale
  Baseline - Youth | 25.15 (6.42) | 24.63 (6.38)
  2 months - Youth | 23.04 (6.43) | 21.59 (6.87)
  4 months - Youth | 21.98 (6.27) | 22.69 (7.04)
  6 months - Youth | 21.34 (6.81) | 21.15 (6.25)
  9 months - Youth | 21.38 (6.76) | 23.28 (7.3)
  12 months - Youth | 22.46 (7.5) | 22.46 (7.02)
Statistical Analysis 1: Comparison: Standard Contingency Management (CM) vs Enhanced Contingency Management (CM+); Mixed effects regression model tested for between-group differences in change over time; Test type: Superiority; p = 0.03, Mixed Models Analysis; Slope = 0.32, Standard Error of Mean 0.15

10. Secondary Outcome: Changes From Baseline Scores Compared to Post-Treatment Scores for Youth Substance Use Frequency (Measured at 0, 2, 4, 6, 9, & 12 Months).
Description: Frequency of substance use as measured by the Global Appraisal of Individual Needs (youth-report).
  The Global Appraisal of Individual Needs (GAIN) Frequency Subscale measures the frequency of substance use of 16 different substances over the past 30 days. Scores range from 0 to 100, where higher scores indicate higher frequency of use.
Time Frame: Baseline to 12 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Standard Contingency Management (CM) | Enhanced Contingency Management (CM+)
Number analyzed (Participants) | 66 | 63
score on a scale
  Baseline | 22.89 (17.37) | 21.9 (17.42)
  2 months | 13.05 (16.09) | 14.51 (15.88)
  4 months | 12.18 (16.94) | 10.48 (15.04)
  6 months | 11.89 (15.11) | 11.15 (12.44)
  9 months | 12.85 (15.63) | 8.06 (14.43)
  12 months | 13.83 (18.76) | 7.51 (11.88)
Statistical Analysis 1: Comparison: Standard Contingency Management (CM) vs Enhanced Contingency Management (CM+); GAIN - Substance Frequency Mixed effects regression model tested for between-group differences in change over time; Test type: Superiority; p = 0.54, Mixed Models Analysis; Slope = -0.21, Standard Error of Mean 0.33

11. Secondary Outcome: Changes From Baseline Scores Compared to Post-Treatment Scores for Youth Substance Problems (Measured at 0, 2, 4, 6, 9, & 12 Months).
Description: The Global Appraisal of Individual Needs (GAIN) Substance Problems Subscale measures the presence of each DSM-V criterion for a substance use disorder and lower severity symptoms. Scores range from 0 to 16, where higher scores indicate the presence of more criterion/symptoms.
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Contingency Management (CM) | Enhanced Contingency Management (CM+)
Number analyzed (Participants) | 66 | 63
score on a scale
  Baseline | 6.73 (4.33) | 7.19 (4.73)
  2 months | 3.91 (3.94) | 3.28 (3.79)
  4 months | 3.33 (3.89) | 2.06 (3.17)
  6 months | 2.51 (3.17) | 2.88 (3.73)
  9 months | 3.14 (3.87) | 1.59 (2.93)
  12 months | 1.95 (2.79) | 1.43 (2.36)
Statistical Analysis 1: Comparison: Standard Contingency Management (CM) vs Enhanced Contingency Management (CM+); Mixed effects regression model tested for between-group differences in change over time; Test type: Superiority; p = 0.89, Mixed Models Analysis; Slope = -0.01, Standard Error of Mean 0.09

12. Secondary Outcome: Changes From Baseline Scores Compared to Post-Treatment Scores for Youth Behavioral Regulation - Risk Taking - Drive - Youth Report (Measured at 0, 2, 4, 6, 9, & 12 Months).
Description: Behavioral regulation - risk taking as measured by the Behavioral Inhibition System and Behavioral Activation System (youth report) scales.
  Youth report of youth risk-taking as assessed by the sum score on the Drive subscale from the Behavioral Inhibition System and Behavioral Activation System scales. Scores on individual items and subscale range from 1=Strongly agree to 4=Strongly disagree and scores range from 4 to 16. Higher scores equal higher youth behavioral activation (drive).
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Contingency Management (CM) | Enhanced Contingency Management (CM+)
Number analyzed (Participants) | 66 | 63
score on a scale
  Baseline - Youth | 11.3 (2.41) | 11.19 (2.31)
  2 months - Youth | 11.17 (2.12) | 11.02 (2.41)
  4 months - Youth | 11.23 (2.01) | 11.09 (2.43)
  6 months - Youth | 10.8 (2.4) | 10.91 (2.3)
  9 months - Youth | 10.91 (2.34) | 11.16 (2.17)
  12 months - Youth | 11.37 (1.96) | 10.82 (2.14)
Statistical Analysis 1: Comparison: Standard Contingency Management (CM) vs Enhanced Contingency Management (CM+); BISBAS Drive - Youth Report. Mixed effects regression model tested for between-group differences in change over time; Test type: Superiority; p = 0.31, Mixed Models Analysis; Slope = 0.05, Standard Error of Mean 0.05

13. Secondary Outcome: Changes From Baseline Scores Compared to Post-Treatment Scores for Youth Behavioral Regulation - Risk Taking - Fun Seeking - Youth Report (Measured at 0, 2, 4, 6, 9, & 12 Months).
Description: Behavioral regulation - risk taking as measured by the Behavioral Inhibition System and Behavioral Activation System (youth report) scales.
  Youth report of youth risk taking as assessed by the sum score on the Fun Seeking subscale from the Behavioral Inhibition System and Behavioral Activation System scales. Scores on individual items and subscale range from 1=Strongly agree to 4=Strongly disagree and scores range from 4 to 16. Higher scores equal higher youth behavioral activation (fun seeking).
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Contingency Management (CM) | Enhanced Contingency Management (CM+)
Number analyzed (Participants) | 66 | 63
score on a scale
  Baseline - Youth | 11.86 (1.8) | 12.46 (1.92)
  2 months - Youth | 12.04 (2.03) | 12.15 (1.98)
  4 months - Youth | 12.03 (2.02) | 12.31 (1.75)
  6 months - Youth | 11.57 (2.4) | 12.41 (1.99)
  9 months - Youth | 11.97 (2.28) | 12.34 (1.54)
  12 months - Youth | 12.03 (1.5) | 12.53 (1.94)
Statistical Analysis 1: Comparison: Standard Contingency Management (CM) vs Enhanced Contingency Management (CM+); Mixed effects regression model tested for between-group differences in change over time; Test type: Superiority; p = 0.35, Mixed Models Analysis; Slope = 0.04, Standard Error of Mean 0.05

14. Secondary Outcome: Changes From Baseline Scores Compared to Post-Treatment Scores for Youth Behavioral Regulation - Risk Taking - Reward Responsiveness - Youth Report (Measured at 0, 2, 4, 6, 9, & 12 Months).
Description: Behavioral regulation - risk taking as measured by the Behavioral Inhibition System and Behavioral Activation System (youth report) scales.
  Youth report of youth risk taking as assessed by the sum score on the Reward Responsiveness subscale from the Behavioral Inhibition System and Behavioral Activation System. Scores on individual items and subscale range from 1=Strongly agree to 4=Strongly disagree and scores range from 5 to 20. Higher scores equal higher youth behavioral activation (reward responsiveness).
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Contingency Management (CM) | Enhanced Contingency Management (CM+)
Number analyzed (Participants) | 66 | 63
score on a scale
  Baseline - Youth | 15.35 (2.43) | 15.41 (2.32)
  2 months - Youth | 15.63 (2.38) | 15.26 (1.95)
  4 months - Youth | 15.48 (2.24) | 15.69 (1.97)
  6 months - Youth | 14.51 (3.02) | 15.44 (1.89)
  9 months - Youth | 15.2 (2.68) | 15.88 (1.81)
  12 months - Youth | 15.63 (2.05) | 15.23 (1.47)
Statistical Analysis 1: Comparison: Standard Contingency Management (CM) vs Enhanced Contingency Management (CM+); Mixed effects regression model tested for between-group differences in change over time; Test type: Superiority; p = 0.13, Mixed Models Analysis; Slope = 0.08, Standard Error of Mean 0.05

15. Secondary Outcome: Changes From Baseline Scores Compared to Post-Treatment Scores for Youth Behavioral Regulation - Risk Taking - Drive - Parent Report (Measured at 0, 2, 4, 6, 9, & 12 Months).
Description: Behavioral regulation - risk taking as measured by the Behavioral Inhibition System and Behavioral Activation System (parent report) scales.
  Parent report of youth risk-taking as assessed by the sum score on the Drive subscale from the Behavioral Inhibition System and Behavioral Activation System scales. Scores on individual items and subscale range from 1=Strongly agree to 4=Strongly disagree and scores range from 4 to 16. Higher scores equal higher youth behavioral activation (drive).
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Contingency Management (CM) | Enhanced Contingency Management (CM+)
Number analyzed (Participants) | 66 | 63
score on a scale
  Baseline - Parent | 11.19 (2.05) | 11.44 (2.6)
  2 months - Parent | 11.92 (2.5) | 11.4 (2.53)
  4 months - Parent | 11.93 (2.87) | 11.48 (2.77)
  6 months - Parent | 12.02 (2.59) | 11.51 (2.75)
  9 months - Parent | 12.05 (2.26) | 11.64 (2.48)
  12 months - Parent | 12.09 (1.91) | 11.19 (2.42)
Statistical Analysis 1: Comparison: Standard Contingency Management (CM) vs Enhanced Contingency Management (CM+); Mixed effects regression model tested for between-group differences in change over time; Test type: Superiority; p = 0.30, Mixed Models Analysis; Slope = -0.04, Standard Error of Mean 0.04

16. Secondary Outcome: Changes From Baseline Scores Compared to Post-Treatment Scores for Youth Behavioral Regulation - Risk Taking - Fun Seeking - Parent Report (Measured at 0, 2, 4, 6, 9, & 12 Months).
Description: Behavioral regulation - risk taking as measured by the Behavioral Inhibition System and Behavioral Activation System (parent report) scales.
  Parent report of youth risk taking as assessed by the sum score on the Fun Seeking subscale from the Behavioral Inhibition System and Behavioral Activation System scales. Scores on individual items and subscale range from 1=Strongly agree to 4=Strongly disagree and scores range from 4 to 16. Higher scores equal higher youth behavioral activation (fun seeking).
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Contingency Management (CM) | Enhanced Contingency Management (CM+)
Number analyzed (Participants) | 66 | 63
score on a scale
  Baseline - Parent | 12.00 (1.72) | 11.84 (1.95)
  2 months - Parent | 11.8 (2.12) | 11.54 (2.16)
  4 months - Parent | 12.16 (2.01) | 11.86 (2.21)
  6 months - Parent | 12.38 (1.85) | 11.49 (2.15)
  9 months - Parent | 12.45 (2.12) | 11.64 (1.78)
  12 months - Parent | 11.93 (2.16) | 11.64 (1.76)
Statistical Analysis 1: Comparison: Standard Contingency Management (CM) vs Enhanced Contingency Management (CM+); Mixed effects regression model tested for between-group differences in change over time; Test type: Superiority; p = 0.70, Mixed Models Analysis; Slope = -0.01, Standard Error of Mean 0.04

17. Secondary Outcome: Changes From Baseline Scores Compared to Post-Treatment Scores for Youth Behavioral Regulation - Risk Taking - Reward Responsiveness - Parent Report (Measured at 0, 2, 4, 6, 9, & 12 Months).
Description: Behavioral regulation - risk taking as measured by the Behavioral Inhibition System and Behavioral Activation System (parent report) scales.
  Parent report of youth risk-taking as assessed by the sum score on the Reward Responsiveness subscale from the Behavioral Inhibition System and Behavioral Activation System. Scores on individual items and subscale range from 1=Strongly agree to 4=Strongly disagree and scores range from 5 to 20. Higher scores equal higher youth behavioral activation (reward responsiveness).
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Contingency Management (CM) | Enhanced Contingency Management (CM+)
Number analyzed (Participants) | 66 | 63
score on a scale
  Baseline - Parent | 15.47 (2.19) | 15.03 (2.36)
  2 months - Parent | 15.29 (2.05) | 15.31 (1.8)
  4 months - Parent | 15.8 (2.08) | 15.09 (2.12)
  6 months - Parent | 15.98 (2.14) | 15.34 (2.08)
  9 months - Parent | 16.1 (2.21) | 15.13 (2.03)
  12 months - Parent | 15.55 (2.26) | 15.62 (1.91)
Statistical Analysis 1: Comparison: Standard Contingency Management (CM) vs Enhanced Contingency Management (CM+); Mixed effects regression model tested for between-group differences in change over time; Test type: Superiority; p = 0.89, Mixed Models Analysis; Slope = 0.01, Standard Error of Mean 0.04

18. Secondary Outcome: Changes From Baseline Scores Compared to Post-Treatment Scores for Youth Behavioral Regulation - Risk Taking - BART (Measured at 0, 2, 4, 6, 9, & 12 Months).
Description: Youth performance on computerized Balloon Analogue Risk Task (automatic version) that requires participants to enter the number of times that they want to pump to inflate a computer-generated balloon, with participants earning a point for each pump but losing all of the points if the balloon pops before the selected number of pumps. The mean number of pumps on all trials is reported. Scores range from 0 to 126. Higher scores equal higher youth risk taking behavior.
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: pumps
Arm/Group | Standard Contingency Management (CM) | Enhanced Contingency Management (CM+)
Number analyzed (Participants) | 66 | 63
pumps
  Baseline | 48.49 (12.17) | 51.72 (13.33)
  2 months | 51.29 (10.3) | 53.86 (11.41)
  4 months | 49.88 (11.85) | 53.14 (11.71)
  6 months | 48.35 (10.37) | 56.29 (14.46)
  9 months | 54.02 (14.9) | 53.90 (13.13)
  12 months | 49.75 (13.67) | 52.09 (13.92)
Statistical Analysis 1: Comparison: Standard Contingency Management (CM) vs Enhanced Contingency Management (CM+); Mixed effects regression model tested for between-group differences in change over time; Test type: Superiority; p = 0.06, Mixed Models Analysis; Slope = -0.50, Standard Error of Mean 0.27

19. Secondary Outcome: Changes From Baseline Scores Compared to Post-Treatment Scores for Youth Behavioral Regulation - Inhibitory Control - EATQ - Youth (Measured at 0, 2, 4, 6, 9, & 12 Months).
Description: Behavioral regulation - inhibitory control as measured by the Early Adolescent Temperament Questionnaire-Revised (youth- and parent-report) and the Go/No Go Task.
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Contingency Management (CM) | Enhanced Contingency Management (CM+)
Number analyzed (Participants) | 66 | 63
score on a scale
  Baseline - Youth | 2.96 (0.63) | 2.8 (0.53)
  2 months - Youth | 3.0 (0.47) | 2.92 (0.57)
  4 months - Youth | 3.01 (0.56) | 3.0 (0.52)
  6 months - Youth | 3.04 (0.48) | 3.06 (0.56)
  9 months - Youth | 3.12 (0.56) | 3.07 (0.45)
  12 months - Youth | 3.17 (0.56) | 3.03 (0.50)
Statistical Analysis 1: Comparison: Standard Contingency Management (CM) vs Enhanced Contingency Management (CM+); EATQ Effortful Control - Youth Report Mixed effects regression model tested for between-group differences in change over time; Test type: Superiority; p = 0.11, Mixed Models Analysis; Slope = -0.02, Standard Error of Mean 0.01

20. Secondary Outcome: Changes From Baseline Scores Compared to Post-Treatment Scores for Youth Behavioral Regulation - Inhibitory Control - EATQ - Parent Report (Measured at 0, 2, 4, 6, 9, & 12 Months).
Description: Parent report of youth inhibitory control as assessed by the mean score on the Effortful Control factor from the Early Adolescent Temperament Questionnaire. Scores on individual items and factor range from 1=Very false to 5=Very true. Higher scores equal higher youth effortful control.
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Contingency Management (CM) | Enhanced Contingency Management (CM+)
Number analyzed (Participants) | 66 | 63
score on a scale
  Baseline - Parent | 2.4 (0.6) | 2.44 (0.54)
  2 months - Parent | 2.47 (0.62) | 2.54 (0.56)
  4 months - Parent | 2.45 (0.59) | 2.55 (0.60)
  6 months - Parent | 2.38 (0.59) | 2.59 (0.59)
  9 months - Parent | 2.42 (0.6) | 2.68 (0.66)
  12 months - Parent | 2.48 (0.61) | 2.73 (0.72)
Statistical Analysis 1: Comparison: Standard Contingency Management (CM) vs Enhanced Contingency Management (CM+); Mixed effects regression model tested for between-group differences in change over time; Test type: Superiority; p = 0.99, Mixed Models Analysis; Slope = -0.0001, Standard Error of Mean 0.009

21. Secondary Outcome: Changes From Baseline Scores Compared to Post-Treatment Scores for Youth Behavioral Regulation - Inhibitory Control - Go No Go Performance (Measured at 0, 2, 4, 6, 9, & 12 Months).
Description: Youth performance of youth inhibitory control as assessed by the percent correct on no go trials on computerized go/no-go task.
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: percent correct
Arm/Group | Standard Contingency Management (CM) | Enhanced Contingency Management (CM+)
Number analyzed (Participants) | 66 | 63
percent correct
  Baseline | 0.74 (0.15) | 0.74 (0.15)
  2 months | 0.75 (0.15) | 0.71 (0.16)
  4 months | 0.73 (0.14) | 0.73 (0.15)
  6 months | 0.75 (0.14) | 0.72 (0.17)
  9 months | 0.77 (0.13) | 0.75 (0.14)
  12 months | 0.73 (0.15) | 0.76 (0.11)
Statistical Analysis 1: Comparison: Standard Contingency Management (CM) vs Enhanced Contingency Management (CM+); Mixed effects regression model tested for between-group differences in change over time; Test type: Superiority; p = 0.82, Mixed Models Analysis; Slope = -0.0007, Standard Error of Mean 0.003

22. Secondary Outcome: Changes From Baseline Scores Compared to Post-Treatment Scores for Peer Relations - Peer Delinquency (Measured at 0, 2, 4, 6, 9, & 12 Months).
Description: Peer relations (association with peers who engage in delinquent behaviors & prosocial activities) as measured by the Peer Relations Questionnaire (youth- and parent-report).
Time Frame: Baseline to 12 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Standard Contingency Management (CM) | Enhanced Contingency Management (CM+)
Number analyzed (Participants) | 66 | 63
score on a scale
  Baseline | 15.42 (13.75) | 14.83 (10.74)
  2 months | 9.89 (9.44) | 10.06 (10.97)
  4 months | 9.38 (9.8) | 11.41 (14.28)
  6 months | 8.8 (8.29) | 8.88 (10.38)
  9 months | 8.06 (7.59) | 9.91 (11.75)
  12 months | 9.45 (12.56) | 7.43 (8.71)
Statistical Analysis 1: Comparison: Standard Contingency Management (CM) vs Enhanced Contingency Management (CM+); Peer Delinquency; Test type: Superiority; p = 0.23, Mixed Models Analysis; Slope = 0.25, Standard Error of Mean 0.21

23. Secondary Outcome: Changes From Baseline Scores Compared to Post-Treatment Scores for Peer Relations - Positive Peer Activity - Youth Report (Measured at 0, 2, 4, 6, 9, & 12 Months).
Description: The Positive Peer Activity Scale of the Pittsburgh Youth Study Interview comprises 10 questions rated on a 4-point scale (0 = none to 4 = all) concerning the proportion of friends of the subject that have engaged in a variety of prosocial activities over the past 30 days. Scores range from 0 to 40, where higher scores indicate a higher proportion of prosocial friends. This is measured from the youth's self-report.
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Contingency Management (CM) | Enhanced Contingency Management (CM+)
Number analyzed (Participants) | 66 | 63
score on a scale
  Baseline - Youth | 16.62 (5.92) | 15.16 (5.94)
  2 months - Youth | 17.37 (6.02) | 16.0 (5.63)
  4 months - Youth | 17.2 (6.01) | 16.28 (7.12)
  6 months - Youth | 17.11 (5.66) | 16.76 (6.16)
  9 months - Youth | 16.66 (5.95) | 18.19 (7.38)
  12 months - Youth | 17.97 (6.5) | 15.71 (5.51)
Statistical Analysis 1: Comparison: Standard Contingency Management (CM) vs Enhanced Contingency Management (CM+); Mixed effects regression model tested for between-group differences in change over time; Test type: Superiority; p = 0.73, Mixed Models Analysis; Slope = 0.04, Standard Error of Mean 0.13

24. Secondary Outcome: Changes From Baseline Scores Compared to Post-Treatment Scores for Peer Relations - Positive Peer Activity - Parent Report (Measured at 0, 2, 4, 6, 9, & 12 Months).
Description: The Positive Peer Activity Scale of the Pittsburgh Youth Study Interview comprises 10 questions rated on a 4-point scale (0 = none to 4 = all) concerning the proportion of friends of the subject that have engaged in a variety of prosocial activities over the past 30 days. Scores range from 0 to 40, where higher scores indicate a higher proportion of prosocial friends. This is measured from the parent's report on youth's friends.
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Contingency Management (CM) | Enhanced Contingency Management (CM+)
Number analyzed (Participants) | 66 | 63
score on a scale
  Baseline - Parent | 9.8 (5.29) | 10.51 (6.56)
  2 months - Parent | 10.41 (5.22) | 11.4 (8.19)
  4 months - Parent | 11.14 (6.04) | 11.0 (7.4)
  6 months - Parent | 10.88 (5.65) | 12.24 (7.02)
  9 months - Parent | 11.4 (4.4) | 13.90 (8.85)
  12 months - Parent | 12.18 (7.15) | 14.39 (7.4)
Statistical Analysis 1: Comparison: Standard Contingency Management (CM) vs Enhanced Contingency Management (CM+); Mixed effects regression model tested for between-group differences in change over time; Test type: Superiority; p = 0.31, Mixed Models Analysis; Slope = 0.11, Standard Error of Mean 0.11

ADVERSE EVENTS:
Time Frame: 1 year post-baseline for each participant.
Arm/Group | Standard Contingency Management (CM) | Enhanced Contingency Management (CM+)
All-Cause Mortality (participants affected / at risk) | 3/66 | 0/63
Serious Adverse Events (participants affected / at risk) | 7/66 | 7/63
Other Adverse Events (participants affected / at risk) | 7/66 | 5/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Contingency Management (CM) (N=66) | Enhanced Contingency Management (CM+) (N=63)
Psychiatric Facility Admission (Psychiatric disorders) | 1 (1) | 1 (1)
Non-fatal Substance Use Overdose (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Suicide Attempt (Psychiatric disorders) | 1 (1) | 2 (2)
Behavioral Escalation (Psychiatric disorders) | 0 (0) | 1 (1)
Physical Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Contingency Management (CM) (N=66) | Enhanced Contingency Management (CM+) (N=63)
Mandatory Child Abuse Report (Social circumstances) | 6 (6) | 5 (5)
Mandatory Report to Law Enforcement (Social circumstances) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/50/NCT03249350/Prot_SAP_000.pdf